CLINICAL TRIAL: NCT06504251
Title: Validity and Reliability of the Modified Delirium Diagnostic Tool - Provisional (DDT-Pro) (Thai Version) in Peri-operative Fragility Hip Fracture Patient
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: COA no. Si 353/2022
Record Dates: First submitted 2024-03-13; First posted 2024-07-16 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2024-07

CONDITIONS: Old Age; Hip Fractures; Delirium
MeSH Terms: conditions — Hip Fractures; Delirium

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Delirium Diagnostic Tool-Provisional ( DDT-Pro ) — The Delirium Diagnostic Tool-Provisional (DDT-Pro) is another tool created to assist in the diagnosis of delirium. It does not require specialist expertise. It can assess the main symptoms of acute confusion, including cognitive ability (Cognition), higher-level thinking skills (Higher level thinking), and the sleep-wake cycle (Sleep-wake cycle).

SUMMARY:
Nowadays, the number of hip fracture patients is increasing. As Thailand enters into an aging society, hip fractures are becoming more common. They are typically treated with surgery. Complications, such as urinary tract infections, pressure sores, and acute confusion, are often observed. These various complications contribute to an increased rate of illness and death.

Delirium is a common problem among hip fracture patients. Currently, diagnosis is typically made using the Diagnostic and Statistical Manual of Mental Disorders (DSM-V), which is a standard tool. However, utilizing it effectively requires expertise. Additionally, other tools such as the Confusion Assessment Method (CAM) and the Memorial Delirium Assessment Scale (MDAS) are available. Nonetheless, training is necessary for their proper use, and they may be more suitable for specific patient groups.

The Delirium Diagnostic Tool-Provisional (DDT-Pro) is another tool created to aid in diagnosing delirium. Unlike other tools, it does not require specialized training. It can assess the main symptoms of delirium, including cognitive ability, higher-level thinking skills, and the sleep-wake cycle. This tool has been utilized in foreign countries such as Spain. The tool was found to have good accuracy and reliability and is useful in aiding the diagnosis of delirium. However, it has never been translated and tested for use in elderly Thai patients with fragility hip fractures.

DETAILED DESCRIPTION:
Inclusion criteria

* Patients older than 65 years
* Had a hip fracture within 7 days before receiving treatment at Siriraj Hospital
* Received surgical treatment for a hip fracture

Exclusion criteria

* Unable to communicate in Thai
* Was diagnosed with cancer before or during treatment for a hip fracture
* Have a history of schizophrenia
* Patients infected with COVID-19

Primary outcomes include:

Validity: Conducting concurrent validity to examine the relationship between the Thai version of DDT-Pro and the Thai version of DSM-V using the 95% confidence interval (CI) for the AUC statistic.

Reliability: Determining the internal consistency of the tool through Cronbach's Alpha with a 95% confidence level, and assessing inter-rater reliability using the 95% CI for Kappa statistic.

Secondary outcomes include:

Prevalence of delirium in patients undergoing surgery for fragility hip fractures

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 65 years
* Hip fracture within a period of 7 days
* Receiving treatment at Siriraj Hospital and who have undergone surgical treatment for the hip fracture.

Exclusion Criteria:

* Unable to communicate in Thai
* Was diagnosed with cancer before or during treatment for a hip fracture
* Have a history of schizophrenia
* Patients infected with COVID-19

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The main objective of the study is to assess the validity and reliability (DDT-Pro) questionnaire in patients with fragility hip fractures before and after receiving surgical treatment.
  For evaluating the Concurrent validity of the tool:
  1. Concurrent validity (95% Confidence Interval (CI) for the Area Under the Curve (AUC))
     - sample size = 99
  2. For reliability assessment (Reliability) of the tool:
     1. Internal consistency (95% confidence level for Cronbach's Alpha)
        - sample size = 90
     2. Inter-rater reliability (95% confidence interval for Kappa) - sample size = 66
  Therefore, the sample size for analyzing inter-rater reliability is at least 66 cases, the sample size for analyzing internal consistency is at least 90 cases, and the sample size for concurrent validity analysis is at least 99 cases. However, the researcher expected a 10% dropout rate, so a sample size of at least 110 cases was used for the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
To evaluate the accuracy and reliability of the revised Thai language version of the Delirium Diagnostic Tool-Provisional (DDT-Pro). | 3 day
  Accuracy and reliability of the revised Thai language version of the Delirium Diagnostic Tool-Provisional (DDT-Pro) compared with the gold standard tool (DSM V)

SECONDARY OUTCOMES:
The incidence of delirium in patients with fragility hip fractures before and after surgical treatment. | 3 day
  Number of delirium in peri-operative fragility hip fracture in Siriraj hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj hospital, Bangkok, Bangkoknoi, Thailand

IPD SHARING:
Plan to Share IPD: Undecided